CLINICAL TRIAL: NCT06610643
Title: Extended Remdesivir Infusion Combined With Nirmatrelvir/Ritonavir for Persistent SARS-CoV-2 Infection in Immunocompromised Patients
Acronym: SARS-CoV-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Clinical professor,, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202405064MIND
Record Dates: First submitted 2024-09-22; First posted 2024-09-24 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: COVID-19; SARS-CoV-2; Immunocompromised
Keywords: Extended RDV infusion combination therapy for SARS-CoV-2 infection in immunocompromised patients
MeSH Terms: conditions — COVID-19 | interventions — Combined Modality Therapy; remdesivir; nirmatrelvir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combination therapy (Experimental): combination of 5-day remdesivir and 10-day Nirmatrelvir/Ritonavir
  Interventions: Drug: combination therapy; Drug: SOC
- SOC (Active Comparator): standard of care
  Interventions: Drug: SOC

INTERVENTIONS:
Drug: combination therapy — A combination of 5-day remdesivir and 10-day Nirmatrelvir/Ritonavir
  Other Names: remdesivir and Nirmatrelvir/Ritonavir
  Arms: combination therapy
Drug: SOC — Standard of care

SUMMARY:
To evaluate the safety and efficacy of extended remdesivir infusion, targeting on immunocompromised individuals who had positive SARS-CoV-2 PCR despite an oral antiviral agent prescription.

DETAILED DESCRIPTION:
Prolonged viral shedding is commonly observed in immunocompromised patients infected by SARS-CoV-2. Until now, there is no successful clinical trial or guideline to guide optimal treatment for this clinical condition. Here, we aimed to establish a clinical trial with combination of prolonged remdesivir infusion with nirmatrelvir/ritonavir among COVID-19 patients recently receiving b-cell depletion therapy, to evaluate to clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Receive B-cell depletion therapy or bendamustine within 6months
* Laboratory confirmed SARS-CoV-2 infection
* Symptoms onset within 72 hours
* NIAID ordinal score 0-5 upon enrollment

Exclusion Criteria:

* Prior use of any anti-SARS-CoV-2 agents within 2 weeks. Remdesivir or NMV/r initiated within 24 hours is acceptable
* Life expectancy < 1 month
* Previous adverse effect related to remdesivir or NMV/r
* Concurrent use medicine with drug-drug interaction with NMV/r
* Patients receiving intubation and mechanical ventilation
* eGFR < 30
* Child pugh score Class C
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-21 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of SARS-CoV-2 CT > 30 on Day 14 | From enrollment to the end of treatment on Day 14.
  The proportion of SARS-CoV-2 CT > 30 on Day 14 of each group.

SECONDARY OUTCOMES:
The proportion of mortality or respiratory failure requiring intubation and mechanical ventilation. | From enrollment to the end of treatment on Day 28.
  The proportion of mortality or respiratory failure requiring intubation and mechanical ventilation within 28 days after antiviral agent initiation of each group.
The proportion of patients developing anti-viral treatment emerging adverse events. | From enrollment to the end of treatment on Day 28.
  The proportion of patients developing anti-viral treatment emerging adverse events.
The proportion of secondary bacterial or fungal infection of each group. | From enrollment to the end of treatment on Day 28.
  The proportion of secondary bacterial or fungal infection of each group.
The proportion of viral rebound within 28 days after antiviral agent initiation. | From enrollment to the end of treatment on Day 28.
  The proportion of viral rebound within 28 days after antiviral agent initiation of each group.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided